CLINICAL TRIAL: NCT03850925
Title: Comparison of Picosecond Pulsed Nd:YAG Laser and Fractional Laser for the Treatment of Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongtan Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Gyeong-Hun Park, Associate professor, Dongtan Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019_02_004
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Acne Scars
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Split-face comparison study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Picosecond laser (Experimental): Intervention: four consecutive sessions of 1,064-nm picosecond laser at 3-week intervals
  Interventions: Procedure: Laser therapy
- Fractional laser (Active Comparator): Intervention: four consecutive sessions of nonablative fractional laser at 3-week intervals
  Interventions: Procedure: Laser therapy

INTERVENTIONS:
Procedure: Laser therapy — 4 consecutive sessions of laser therapy

SUMMARY:
This study compares the application of a picosecond 1064-nm laser with a diffractive lens array with nonablative fractional laser for the treatment of acne scarring.

DETAILED DESCRIPTION:
This trial is a 17-week, prospective, randomized split-face study that compares the results between two facial sides either receiving the picosecond 1064-nm laser or nonablative fractional laser treatment for atrophic acne scar.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with facial atrophic acne scars
* Subjects who observe the schedules and protocols of the clinical trial
* Subjects who give informed consent to participate in the clinical trial

Exclusion Criteria:

* Subjects who have active acne under treatment
* Subjects who had received any other treatments for acne scarring for 6 months prior to the first treatment
* Subjects who underwent other treatments including chemical, mechanical or laser resurfacing during the study period
* Subjects who have current acute illness
* Subjects who are considered inappropriate for the clinical trial under the judgement of investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the mean of the ECCA grading scale | Week 17
  The ECCA (échelle d'évaluation clinique des cicatrices d'acné) grading scale: minimum score 0; maximum score 270; higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gyeong-Hun Park, MD, PhD, Principal Investigator — Dongtan Sacred Heart Hospital, Hallym University College of Medicine
Locations (1):
- Dongtan Sacred Heart Hospital, Hallym Universtiy College of Medicine, Hwaseong-si, Gyeonggi-do, South Korea